CLINICAL TRIAL: NCT01370993
Title: The Prediction Model of Hypoxemia for Safe Bronchoscopy Under MAC Anesthesia
Brief Title: The Prediction Model of Hypoxemia for Safe Bronchoscopy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Sei Won Lee/Assistant professor, Seoul National University Bundang Hospital
Other Study IDs: SNUBH-FOB under MAC
Record Dates: First submitted 2011-05-31; First posted 2011-06-10 (Estimated); Last update posted 2011-06-10 (Estimated); Status verified 2011-05

CONDITIONS: Hypoxemia; Obstructive Sleep Apnea
Keywords: Hypoxemia; Model; Bronchoscopes; Monitored anesthesia care
MeSH Terms: conditions — Hypoxia; Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to develop the hypoxemia prediction model during fiberoptic bronchoscopy under MAC(monitored anesthesia care) anesthesia.

DETAILED DESCRIPTION:
Currently, diverse sedatives and analgesic methods are used during fiberoptic bronchoscopy for reducing patients' discomfort and facilities of procedures as British Thoracic Society recommendation. MAC anesthesia, one of the widely used sedative method during bronchoscopy, have many advantages, occurrence of respiratory depression, hypoxemia are not uncommon during the procedures. The investigators try to find out risk factors and develop the prediction model for hypoxemia during bronchoscopy under MAC anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Age> 15 yrs
* patients who are planned to get fiberoptic bronchoscopy under MAC anesthesia in Seoul National University Bundang Hospital

Exclusion Criteria:

* Patients who will get Endobronchial ultrasound guided transbronchial needle aspiration
* patients whose baseline oxygen saturation is below 90%
* Intubated patients
* Patients do not agree with the study enrollment

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patienst who are planned to get fiberoptic bronchoscopy under MAC anesthesia in Seoul National University Bundang Hospital
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2011-05; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Lowest oxygen saturation during bronchoscopy, development of hypoxemia(SpO2<90%) during bronchoscopy | during the fiberoptic bronchoscopy, estimated procedure time is about 15min

SECONDARY OUTCOMES:
Need for oxygen flow increment | during the fiberoptic bronchoscopy, estimated procedure time is about 15min
the proportion of subjects who is require of mandible lift | during the fiberoptic bronchoscopy, estimated procedure time is about 15min
time delay for procedure due to hypoxemia | during the fiberoptic bronchoscopy, estimated procedure time is about 15min
the proportion of subjects with snoring | during the fiberoptic bronchoscopy, estimated procedure time is about 15min
  snoring

CONTACTS AND LOCATIONS:
Overall Officials: Sei Won Lee, M.D., Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Sei Won Lee, Seongnam-si, Gyeonggi-do, South Korea